CLINICAL TRIAL: NCT05498298
Title: A Cross-sectional, Interventional, Exploratory Clinical Study to Investigate the Reliability of Fetal Heart Rate and Maternal Heart Rate Signals Extracted From Biopotential Data
Brief Title: A Clinical Study to Investigate the Reliability of Fetal Heart Rate and Maternal Heart Rate Signals Extracted From Biopotential Data
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bloom Technologies (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: LOV-02-2022-US
Record Dates: First submitted 2022-08-09; First posted 2022-08-12 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Pregnancy Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Gtec (Experimental)
  Interventions: Device: Biopotentials measurement with gtec device

INTERVENTIONS:
Device: Biopotentials measurement with gtec device — A measurement of 40 minutes is performed with the gtec g.Hlamp to collect biopotential signals. 32 electrodes are attached to the body (abdomen, thorax and back).

SUMMARY:
Bloom Technologies is developing a wearable device for monitoring pregnancy.

In this study, Bloom Technologies wants to investigate the reliability of this new technology.

For this reason, a device that records very high-quality data (g,Hlamp) was chosen. The study device is attached to the body by means of electrodes (up to 32) that can be safely attached to the skin. Most of the electrodes are placed on the abdomen, and a few on the chest and back.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant woman ≥ 18 years old
* Gestational age ≥ 30 weeks and 0 days
* Singleton pregnancy
* Ability to read and understand English or Spanish
* Willingness to participate in the study

Exclusion Criteria:

* Implanted pacemaker or any other implanted electrical device
* History of allergies to skin adhesives
* Irritated or lesioned skin at the electrodes locations

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2022-12-07 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Reliability in fetal heart rate extraction | 40 minutes
  Percentage of a recording with a fetal heart rate signal extracted
Reliability in maternal heart rate extraction | 40 minutes
  Percentage of a recording with a maternal heart rate signal extracted

CONTACTS AND LOCATIONS:
Overall Officials: Ravindu Gunatilake, Principal Investigator — Valley Perinatal Services
Locations (1):
- Valley Perinatal Services, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided